CLINICAL TRIAL: NCT01447355
Title: Pilot Study on the Bioactivity of Vitamin D in the Skin After Oral Supplementation
Brief Title: Vitamin D Levels in the Skin of Healthy Subjects After Oral Supplementation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2011-03469; NCI-2011-03469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000712963; 11-0270-04 (Other: University of Arizona Health Sciences Center); UAZ10-16-03 (Other: DCP); N01CN35158 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Healthy, no Evidence of Disease; Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Cholecalciferol

ARMS (1):
- Prevention (cholecalciferol) (Experimental): Participants receive cholecalciferol PO twice weekly for up to 8-9 weeks.
  Interventions: Drug: cholecalciferol

INTERVENTIONS:
Drug: cholecalciferol — Given PO
  Other Names: Calciol; Vitamin D3

SUMMARY:
This pilot phase I trial studies vitamin D levels in the skin of healthy subjects after oral supplementation. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of cholecalciferol, a vitamin D, may keep skin cancer from forming.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if high-dose oral cholecalciferol supplementation increases vitamin D receptor (VDR) expression in keratinocytes from photoprotected areas in healthy subjects with documented insufficient serum levels of 25-hydroxyvitamin D (defined as =< 30.0 ng/mL).

SECONDARY OBJECTIVES:

I. To assess the modulation in CYP24 expression in keratinocytes (from photoprotected and photodamaged skin samples).

II. To assess the modulation in VDR expression in keratinocytes (from photodamaged skin samples).

III. To assess the mechanistic information concerning the action of cholecalciferol supplementation in the state of keratinocytic differentiation by assessing caspase 14, loricrin, and assessment of stratum corneum thickness.

IV. To assess the safety and tolerability of high-dose cholecalciferol supplementation in this patient cohort, including the evaluation of calcium, phosphate, and parathyroid hormone (PTH).

V. To assess the 25-hydroxyvitamin D levels after intervention supplementation.

TERTIARY OBJECTIVES:

I. To assess the corresponding VDR and CYP24 expression in benign melanocytic nevi. (Exploratory)

OUTLINE:

Participants receive cholecalciferol orally (PO) twice weekly for up to 8-9 weeks.

After completion of study treatment, participants are followed up for 10-14 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented insufficient serum levels of 25-hydroxyvitamin D =< 30.0 ng/mL
* At least moderate sun-damaged skin on the mid-upper right dorsal forearm
* Karnofsky performance status of at least 80%
* Leukocytes ÃÂ¢ÃÂ¥ 3,000/ÃÃÂ¼L
* Absolute neutrophil count ÃÂ¢ÃÂ¥ 1,500/ÃÃÂ¼L
* Platelets ÃÂ¢ÃÂ¥ 100,000/ÃÃÂ¼L
* Total bilirubin ÃÂ¢ÃÂ¤ 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< institutional upper limit of normal (ULN)
* Creatinine ÃÂ¢ÃÂ¤ 1.4 mg/dL
* Serum calcium 8.4-10.6 mg/dL
* Parathyroid hormone (PTH): male 8.3-10.4 mg/dL; female 8.4-10.6 mg/dL
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence; surgical sterilization; or at least one year post-menopausal) prior to study entry and for the duration of study participation
* Skin phototype II or III as defined according to their skin response to sunlight:

  * Skin phototype II will always burn, and tan minimally after 45-60 min of unprotected exposure to the summer sun between 12-1pm
  * Skin phototype III will sometimes burn, and almost always tan after 45-60 min of unprotected exposure to the summer sun between 12-1pm
* Ability to understand and willingness to sign written informed consent
* Participants may not have acute or chronic hypervitaminosis D or hypercalcemia
* No history of increased arterial calcification or atherosclerosis, sarcoidosis, histoplasmosis, hyperparathyroidism, lymphoma, or kidney disease
* No current use of digoxin (Lanoxin, digitalis), cholestyramine (Prevalite, Questran), colestipol (Cholestid), oral steroids (prednisone and others), and antacids that contain magnesium
* Participants may not be receiving any other investigational agents; if they have completed a clinical-intervention trial recently, there must be a 30-day period between completing the previous study and entering this study
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to cholecalciferol, lidocaine, or xylocaine
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded from this study
* No invasive cancer or cancer treatment within the past five years, except non-melanoma skin cancer
* No immunosuppression by virtue of medication or disease; this includes acquired immune deficiency syndrome (AIDS) patients, subjects taking oral prednisone, and subjects on immunosuppressants/immunomodulators (cyclosporine, chemotherapeutic agents, or biologic therapy), as determined by the examining investigator/co-investigator
* Unwilling or unable to refrain from taking herbal medicines or above-standard vitamin or mineral during the study

  * A standard daily multivitamin/mineral supplement is acceptable if it contains ÃÃÂ¢ÃÃÂ¤ 600 IU of vitamin D, or ÃÃÂ¢ÃÃÂ¤ the recommended dietary allowance (RDA) of calcium, and the subject has been taking a stable dose for at least 30 days
  * Potential subjects who are taking above-standard doses of supplements may be re-considered for participation after a 30-day wash-out period
* No participants who have used tanning beds or other methods to promote sun-tanning within 6 months of study entry; such practices may not be undertaken during participation in the study
* Participants unwilling to minimize their exposure to sunlight by applying sunscreen/sunblock or by wearing clothing to shield their skin, during outdoor activities, while they are enrolled in the study
* Individuals receiving concurrent topical therapy with retinoids, steroids, 5-fluorouracil, Levulan, Vaniqa (eflornithine), Solaraze, or Imiquimod (AldaraÃÃÃÂ®) within 30 days prior to study enrollment will be excluded; subjects may be reconsidered for eligibility 30 days after the last treatment
* Individuals who have had treatment for basal cell carcinoma or squamous cell carcinoma on the skin of the right forearm within six months prior to evaluation for the study will not be eligible; these subjects will be encouraged to return for re-evaluation once the six-month period is over

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in VDR expression from baseline to post-intervention | From baseline to post-intervention

SECONDARY OUTCOMES:
Modulation in CYP24 expression in keratinocytes in photoprotected and photodamaged areas | Up to 9 weeks
Modulation of VDR in keratinocytes in photodamaged skin | Up to 9 weeks
Changes in a panel of biomarkers of skin differentiation including caspase 14, loricrin, and stratum corneum thickness in keratinocytes in photo-protected and damaged skin | From baseline to 9 weeks
Changes in 25-hydroxyvitamin D serum levels | From baseline to 9 weeks
Changes in calcium, phosphate, and PTH | From baseline to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clara Curiel-Lewandrowski, Principal Investigator — University of Arizona Health Sciences Center
Locations (1):
- University of Arizona Health Sciences Center, Tucson, Arizona, United States